CLINICAL TRIAL: NCT02826798
Title: A Phase 1 Randomized, Observer-Blind, Placebo-Controlled, Study to Evaluate the Safety, Tolerability, and Immunogenicity of the Candidate Human Cytomegalovirus Vaccine (VBI-1501) in Healthy Adults
Brief Title: Study to Evaluate Safety, Tolerability, and Immunogenicity of Candidate Human Cytomegalovirus Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VBI Vaccines Inc. (Industry)
Collaborators: Clinical Trial Data Services, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VBI-1501
Record Dates: First submitted 2016-06-23; First posted 2016-07-11 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Cytomegalovirus Infections
Keywords: VBI-1501A; VBI-1501; prophylactic vaccine; virus diseases; cytomegalovirus (CMV); cytomegalovirus infections; cytomegalovirus vaccines; Herpesviridae Infections; Phase 1; Human Herpesvirus 5 (HHV5); Vaccines, virus-like particle (VLP); enveloped virus-like particle (eVLP)
MeSH Terms: conditions — Cytomegalovirus Infections; Virus Diseases; Herpesviridae Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- VBI-1501A: 0.5µg with adjuvant (Experimental): 0.5µg CMV vaccine with adjuvant
  Interventions: Drug: VBI-1501A 0.5 μg
- VBI-1501A: 1.0µg with adjuvant (Experimental): 1.0µg CMV vaccine with adjuvant
  Interventions: Drug: VBI-1501A 1.0 μg
- VBI-1501A: 2.0 µg with adjuvant (Experimental): 2.0 µg CMV vaccine with adjuvant
  Interventions: Drug: VBI-1501A 2.0 μg
- VBI-1501: 1.0µg without adjuvant (Experimental): 1.0µg CMV vaccine without adjuvant
  Interventions: Drug: VBI-1501 1.0 μg
- Placebo (Placebo Comparator): Buffer/sucrose used for VBI-1501 suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VBI-1501A 0.5 μg — VBI-1501A: 0.5 μg with alum-administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
  Arms: VBI-1501A: 0.5µg with adjuvant
Drug: VBI-1501A 1.0 μg — VBI-1501A: 1.0 μg with alum with alum-administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
  Arms: VBI-1501A: 1.0µg with adjuvant
Drug: VBI-1501A 2.0 μg — VBI-1501A: 2.0 μg with alum-administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
  Arms: VBI-1501A: 2.0 µg with adjuvant
Drug: VBI-1501 1.0 μg — VBI-1501: 1.0 μg without alum-administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
  Arms: VBI-1501: 1.0µg without adjuvant
Drug: Placebo — buffer/sucrose used for VBI-1501 suspension- administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of four different doses of cytomegalovirus vaccines in healthy adults.

DETAILED DESCRIPTION:
This study is designed to assess safety and immunogenicity of four dose formulations of cytomegalovirus (CMV) vaccine (0.5 μg gB content with aluminum phosphate (alum), 1.0 μg glycoprotein B (gB) content with alum, 2.0 μg gB content with alum, or 1.0 μg gB content (without alum) as compared with placebo in approximately 125 healthy CMV-seronegative volunteer participants between 18 and 40 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy adult female and male 18 to 40 years of age, inclusive;
2. Serologically confirmed to be CMV seronegative at screening;
3. Female volunteers must agree to use an adequate contraception method as deemed appropriate by the investigator
4. Sign an informed consent document indicating understanding of the purpose and procedures required for the study and willingness to participate in the study

Exclusion Criteria:

1. History of or current clinically significant medical illness or any other illness that in the opinion of the investigator interferes with the interpretation of the study results
2. Clinically significant abnormal physical examination, vital signs, or clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening as determined by the investigator
3. Previous receipt of any cytomegalovirus vaccine
4. History of allergic reactions or anaphylactic reaction to any vaccine component
5. Pregnant or breastfeeding or plans to conceive from two weeks before the study start through six months after the last dose of study vaccine
6. Known or suspected impairment of immunological function, including but not limited to autoimmune diseases, splenectomy, or HIV/AIDS
7. Chronic administration (defined as more than 14 days in total) of immune-suppressive or other immune-modifying drug with six months prior to the product dose (for corticosteroids, this is defined as prednisone ≥20 mg/day or equivalent). Inhaled and topical steroids are allowed
8. Participation in another clinical study within 30 days or plans to participate in another treatment based clinical study during the conduct of the present study
9. Any skin abnormality or tattoo that would limit post-vaccination injection site assessment
10. Any history of cancer requiring chemotherapy or radiation within 5 years of randomization or current disease
11. Are family members of study center staff

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2017-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Langley, MD, Principal Investigator — IWK Health Centre
Locations (3):
- Canada (3):
  - Vaccine Evaluation Center, Vancouver, British Columbia
  - Canadian Center for Vaccinology; IWK Health Centre, Halifax, Nova Scotia
  - McGill University Health Centre - Vaccine Study, Pierrefonds, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler SP, Starr SE, Plotkin SA, Hempfling SH, Buis J, Manning ML, Best AM. Immunity induced by primary human cytomegalovirus infection protects against secondary infection among women of childbearing age. J Infect Dis. 1995 Jan;171(1):26-32. doi: 10.1093/infdis/171.1.26. PMID 7798679
- [Background] Adler SP. Human CMV vaccine trials: what if CMV caused a rash? J Clin Virol. 2008 Mar;41(3):231-6. doi: 10.1016/j.jcv.2007.11.008. Epub 2007 Dec 21. PMID 18096431
- [Background] Axelsson F, Adler SP, Lamarre A, Ohlin M. Humoral immunity targeting site I of antigenic domain 2 of glycoprotein B upon immunization with different cytomegalovirus candidate vaccines. Vaccine. 2007 Dec 21;26(1):41-6. doi: 10.1016/j.vaccine.2007.10.048. Epub 2007 Nov 9. PMID 18063447
- [Background] Baylor NW, Egan W, Richman P. Aluminum salts in vaccines--US perspective. Vaccine. 2002 May 31;20 Suppl 3:S18-23. doi: 10.1016/s0264-410x(02)00166-4. PMID 12184360
- [Background] Biffi A, Montini E, Lorioli L, Cesani M, Fumagalli F, Plati T, Baldoli C, Martino S, Calabria A, Canale S, Benedicenti F, Vallanti G, Biasco L, Leo S, Kabbara N, Zanetti G, Rizzo WB, Mehta NA, Cicalese MP, Casiraghi M, Boelens JJ, Del Carro U, Dow DJ, Schmidt M, Assanelli A, Neduva V, Di Serio C, Stupka E, Gardner J, von Kalle C, Bordignon C, Ciceri F, Rovelli A, Roncarolo MG, Aiuti A, Sessa M, Naldini L. Lentiviral hematopoietic stem cell gene therapy benefits metachromatic leukodystrophy. Science. 2013 Aug 23;341(6148):1233158. doi: 10.1126/science.1233158. Epub 2013 Jul 11. PMID 23845948
- [Background] Amai M, Nojima M, Yuki Y, Kiyono H, Nagamura F. A review of criteria strictness in "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". Vaccine. 2023 Aug 31;41(38):5622-5629. doi: 10.1016/j.vaccine.2023.07.072. Epub 2023 Aug 1. PMID 37532612
- [Background] Fishman JA, Emery V, Freeman R, Pascual M, Rostaing L, Schlitt HJ, Sgarabotto D, Torre-Cisneros J, Uknis ME. Cytomegalovirus in transplantation - challenging the status quo. Clin Transplant. 2007 Mar-Apr;21(2):149-58. doi: 10.1111/j.1399-0012.2006.00618.x. PMID 17425738
- [Background] Fu TM, Wang D, Freed DC, Tang A, Li F, He X, Cole S, Dubey S, Finnefrock AC, ter Meulen J, Shiver JW, Casimiro DR. Restoration of viral epithelial tropism improves immunogenicity in rabbits and rhesus macaques for a whole virion vaccine of human cytomegalovirus. Vaccine. 2012 Dec 14;30(52):7469-74. doi: 10.1016/j.vaccine.2012.10.053. Epub 2012 Oct 26. PMID 23107592
- [Background] Gordon EM, Levy JP, Reed RA, Petchpud WN, Liu L, Wendler CB, Hall FL. Targeting metastatic cancer from the inside: a new generation of targeted gene delivery vectors enables personalized cancer vaccination in situ. Int J Oncol. 2008 Oct;33(4):665-75. PMID 18813779
- [Background] Griffiths PD, Stanton A, McCarrell E, Smith C, Osman M, Harber M, Davenport A, Jones G, Wheeler DC, O'Beirne J, Thorburn D, Patch D, Atkinson CE, Pichon S, Sweny P, Lanzman M, Woodford E, Rothwell E, Old N, Kinyanjui R, Haque T, Atabani S, Luck S, Prideaux S, Milne RS, Emery VC, Burroughs AK. Cytomegalovirus glycoprotein-B vaccine with MF59 adjuvant in transplant recipients: a phase 2 randomised placebo-controlled trial. Lancet. 2011 Apr 9;377(9773):1256-63. doi: 10.1016/S0140-6736(11)60136-0. PMID 21481708
- [Background] Hacein-Bey-Abina S, Pai SY, Gaspar HB, Armant M, Berry CC, Blanche S, Bleesing J, Blondeau J, de Boer H, Buckland KF, Caccavelli L, Cros G, De Oliveira S, Fernandez KS, Guo D, Harris CE, Hopkins G, Lehmann LE, Lim A, London WB, van der Loo JC, Malani N, Male F, Malik P, Marinovic MA, McNicol AM, Moshous D, Neven B, Oleastro M, Picard C, Ritz J, Rivat C, Schambach A, Shaw KL, Sherman EA, Silberstein LE, Six E, Touzot F, Tsytsykova A, Xu-Bayford J, Baum C, Bushman FD, Fischer A, Kohn DB, Filipovich AH, Notarangelo LD, Cavazzana M, Williams DA, Thrasher AJ. A modified gamma-retrovirus vector for X-linked severe combined immunodeficiency. N Engl J Med. 2014 Oct 9;371(15):1407-17. doi: 10.1056/NEJMoa1404588. PMID 25295500
- [Background] Institute of Medicine (US) Committee to Study Priorities for Vaccine Development; Stratton KR, Durch JS, Lawrence RS, editors. Vaccines for the 21st Century: A Tool for Decisionmaking. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK233313/ PMID 25121214
- [Background] Loomis RJ, Lilja AE, Monroe J, Balabanis KA, Brito LA, Palladino G, Franti M, Mandl CW, Barnett SW, Mason PW. Vectored co-delivery of human cytomegalovirus gH and gL proteins elicits potent complement-independent neutralizing antibodies. Vaccine. 2013 Jan 30;31(6):919-26. doi: 10.1016/j.vaccine.2012.12.009. Epub 2012 Dec 14. PMID 23246547
- [Background] Macagno A, Bernasconi NL, Vanzetta F, Dander E, Sarasini A, Revello MG, Gerna G, Sallusto F, Lanzavecchia A. Isolation of human monoclonal antibodies that potently neutralize human cytomegalovirus infection by targeting different epitopes on the gH/gL/UL128-131A complex. J Virol. 2010 Jan;84(2):1005-13. doi: 10.1128/JVI.01809-09. Epub 2009 Nov 4. PMID 19889756
- [Background] 15. Paneque-Quevedo AA. Inorganic compounds as vaccine adjuvants. Biotecnología Aplicada. 2013;30:250-256.
- [Background] Pass RF, Duliege AM, Boppana S, Sekulovich R, Percell S, Britt W, Burke RL. A subunit cytomegalovirus vaccine based on recombinant envelope glycoprotein B and a new adjuvant. J Infect Dis. 1999 Oct;180(4):970-5. doi: 10.1086/315022. PMID 10479120
- [Background] Pass RF, Zhang C, Evans A, Simpson T, Andrews W, Huang ML, Corey L, Hill J, Davis E, Flanigan C, Cloud G. Vaccine prevention of maternal cytomegalovirus infection. N Engl J Med. 2009 Mar 19;360(12):1191-9. doi: 10.1056/NEJMoa0804749. PMID 19297572
- [Background] Plotkin SA. Is there a formula for an effective CMV vaccine? J Clin Virol. 2002 Aug;25 Suppl 2:S13-21. doi: 10.1016/s1386-6532(02)00093-8. No abstract available. PMID 12361753
- [Background] Zydek M, Petitt M, Fang-Hoover J, Adler B, Kauvar LM, Pereira L, Tabata T. HCMV infection of human trophoblast progenitor cells of the placenta is neutralized by a human monoclonal antibody to glycoprotein B and not by antibodies to the pentamer complex. Viruses. 2014 Mar 19;6(3):1346-64. doi: 10.3390/v6031346. PMID 24651029
- [Derived] Langley JM, Gantt S, Halperin SA, Ward B, McNeil S, Ye L, Cai Y, Smith B, Anderson DE, Mitoma FD. An enveloped virus-like particle alum-adjuvanted cytomegalovirus vaccine is safe and immunogenic: A first-in-humans Canadian Immunization Research Network (CIRN) study. Vaccine. 2024 Jan 25;42(3):713-722. doi: 10.1016/j.vaccine.2023.12.019. Epub 2023 Dec 22. PMID 38142214

RESULTS

PARTICIPANT FLOW:
Groups:
- VBI-1501A: 0.5µg With Adjuvant: Healthy cytomegalovirus (CMV)-seronegative subjects between 18 and 40 years of age received three doses of 0.5 μg VBI-1501A human CMV glycoprotein B (gB) adsorbed on Adju-Phos® adjuvant administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
- VBI-1501A: 1.0µg With Adjuvant: Healthy CMV-seronegative subjects between 18 and 40 years of age received three doses of 1.0 μg VBI-1501A human CMV glycoprotein B (gB) adsorbed on Adju-Phos® adjuvant administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
- VBI-1501A: 2.0 µg With Adjuvant: Healthy CMV-seronegative subjects between 18 and 40 years of age received three doses of 2.0 μg VBI-1501A human CMV glycoprotein B (gB) adsorbed on Adju-Phos® adjuvant administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
- VBI-1501: 1.0µg Without Adjuvant: Healthy CMV-seronegative subjects between 18 and 40 years of age received three doses of 1.0 μg VBI-1501 human CMV without adjuvant administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
- Placebo: Healthy CMV-seronegative subjects between 18 and 40 years of age received three doses of buffer/sucrose used for VBI-1501 suspension administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
Period: Overall Study
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
Started | 25 | 26 | 26 | 25 | 26
Completed | 25 | 25 | 26 | 24 | 26
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- VBI-1501A: 0.5µg With Adjuvant: Healthy CMV-seronegative subjects between 18 and 40 years of age received three doses of 0.5 μg VBI-1501A human CMV glycoprotein B (gB) adsorbed on Adju-Phos® adjuvant administered as a 0.5 mL intramuscular injection on Days 0, 56, and 168
- Total: Total of all reporting groups
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo | Total
Number analyzed (Participants) | 25 | 26 | 26 | 25 | 26 | 128
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean (standard deviation) | 26.4 (4.58) | 27.0 (5.38) | 26.5 (4.60) | 26.8 (5.99) | 28.3 (5.58) | 27.0 (5.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 17 | 14 | 15 | 76
  Male | 13 | 8 | 9 | 11 | 11 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  North American Indian | 0 | 0 | 0 | 0 | 0 | 0
  White, Caucasian | 22 | 24 | 23 | 22 | 24 | 115
  Chinese | 2 | 1 | 0 | 1 | 1 | 5
  Black | 0 | 0 | 0 | 1 | 0 | 1
  Filipino | 0 | 1 | 0 | 0 | 0 | 1
  West Asian | 0 | 0 | 1 | 0 | 0 | 1
  Alaskan Native | 0 | 0 | 1 | 0 | 0 | 1
  Other | 1 | 0 | 1 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 26 | 26 | 25 | 26 | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Adverse Events During Seven-Day Follow-Up Period
Time Frame: Day of vaccine administration (days 0, 56, 168) and six subsequent days
Population: Analyses were performed on the total vaccinated cohort (TVC), which includes all immunized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 23 | 26
Participants
  Pain at injection site, Dose 1: number analyzed (Participants) | 25 | 25 | 25 | 22 | 26
  Pain at injection site, Dose 1 | 11 | 14 | 13 | 5 | 3
  Pain at injection site, Dose 2 | 10 | 15 | 14 | 5 | 4
  Pain at injection site, Dose 3: number analyzed (Participants) | 24 | 25 | 25 | 23 | 26
  Pain at injection site, Dose 3 | 10 | 13 | 13 | 4 | 3
  Fatigue, Dose 1: number analyzed (Participants) | 25 | 25 | 25 | 22 | 26
  Fatigue, Dose 1 | 9 | 8 | 5 | 11 | 6
  Fatigue, Dose 2 | 9 | 7 | 8 | 8 | 3
  Fatigue, Dose 3 | 10 | 7 | 7 | 7 | 3
  Diarrhea, Dose 1: number analyzed (Participants) | 25 | 25 | 25 | 22 | 26
  Diarrhea, Dose 1 | 6 | 4 | 2 | 4 | 3
  Diarrhea, Dose 2 | 2 | 3 | 1 | 0 | 1
  Diarrhea, Dose 3 | 2 | 1 | 3 | 2 | 0
  Nausea/Vomiting, Dose 1: number analyzed (Participants) | 25 | 25 | 25 | 22 | 26
  Nausea/Vomiting, Dose 1 | 4 | 2 | 2 | 2 | 1
  Nausea/Vomiting, Dose 2 | 2 | 4 | 4 | 0 | 0
  Nausea/Vomiting, Dose 3 | 1 | 2 | 3 | 0 | 0
  Headache, Dose 1: number analyzed (Participants) | 25 | 25 | 25 | 22 | 26
  Headache, Dose 1 | 9 | 11 | 7 | 10 | 7
  Headache, Dose 2 | 11 | 8 | 10 | 10 | 2
  Headache, Dose 3 | 7 | 12 | 9 | 10 | 5
  Malaise, Dose 1: number analyzed (Participants) | 25 | 25 | 25 | 22 | 26
  Malaise, Dose 1 | 8 | 7 | 4 | 7 | 4
  Malaise, Dose 2 | 5 | 8 | 7 | 3 | 3
  Malaise, Dose 3 | 5 | 6 | 4 | 4 | 2
  Myalgia, Dose 1: number analyzed (Participants) | 25 | 24 | 25 | 22 | 26
  Myalgia, Dose 1 | 6 | 11 | 1 | 4 | 3
  Myalgia, Dose 2 | 2 | 8 | 3 | 3 | 1
  Myalgia, Dose 3 | 4 | 5 | 2 | 1 | 2
  Neck Swelling, Dose 1: number analyzed (Participants) | 25 | 25 | 25 | 22 | 26
  Neck Swelling, Dose 1 | 2 | 3 | 2 | 0 | 3
  Neck Swelling, Dose 2 | 2 | 1 | 1 | 2 | 3
  Neck Swelling, Dose 3 | 1 | 2 | 3 | 2 | 1
  Armpit Swelling, Dose 1: number analyzed (Participants) | 25 | 25 | 25 | 22 | 26
  Armpit Swelling, Dose 1 | 1 | 1 | 1 | 0 | 2
  Armpit Swelling, Dose 2 | 1 | 0 | 0 | 2 | 1
  Armpit Swelling, Dose 3 | 0 | 0 | 0 | 1 | 1

2. Primary Outcome: Number of Participants With Any Adverse Event
Time Frame: Following each of the 3 injections of study vaccine, the occurrence of adverse events was captured during a 28-day follow-up period as well as through Day 336 or early withdrawal.
Population: Analyses were performed on the total vaccinated cohort (TVC), which includes all immunized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 23 | 26
Participants
  Post-Dose 1 | 12 | 11 | 10 | 10 | 15
  Post-Dose 2 | 8 | 11 | 10 | 8 | 8
  Post-Dose 3 | 7 | 13 | 8 | 8 | 7
  Through Day 336 or Early Withdrawal | 18 | 22 | 19 | 19 | 22

3. Primary Outcome: Number of Participants With Any Serious Adverse Event
Time Frame: Through Day 336 or early withdrawal
Population: Analyses were performed on the total vaccinated cohort (TVC), which includes all immunized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 23 | 26
Participants | 0 | 2 | 0 | 2 | 0

4. Primary Outcome: Number of Participants With Any Hematological or Biochemical Laboratory Abnormality
Description: Blood and urine samples were collected at screening for all evaluations with additional blood samples obtained on Days 28, 56, 84, 168, 196, 280, and 336. The following clinical laboratory evaluations were performed: Biochemistry: alanine aminotransferase; aspartate aminotransferase; creatinine; blood urea nitrogen; Hematology: neutrophils, lymphocytes, eosinophils, hemoglobin, platelet count, white blood cell count; Infection status: HIV, hepatitis B, hepatitis C, and cytomegalovirus; and Urinalysis: blood, glucose, protein.
Time Frame: Through Day 336 or early withdrawal
Population: Analyses were performed on the total vaccinated cohort (TVC), which includes all immunized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 23 | 26
Participants
  Day 28 | 14 | 10 | 15 | 8 | 11
  Day 56 | 13 | 13 | 15 | 14 | 11
  Day 84 | 13 | 11 | 13 | 13 | 14
  Day 168 | 16 | 11 | 14 | 13 | 14
  Day 196 | 12 | 13 | 15 | 13 | 11
  Day 280 | 14 | 13 | 13 | 13 | 16
  Day 336 | 14 | 14 | 16 | 13 | 14

5. Secondary Outcome: Geometric Mean Titer of Antibody Binding to CMV gB
Time Frame: Through Day 336 or early withdrawal
Population: Analyses were performed on the total vaccinated cohort (TVC), which includes all immunized subjects. The group means and standard deviations of positive samples are shown, except where no samples tested positive (neither mean nor standard deviation could be calculated) or only one sample tested positive (standard deviation could not be calculated).
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 23 | 26
Titer
  Day 0 | 1126.00 (NA) — Standard deviation not calculated because only one participant's sample measured above the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | 1077.29 (1.85) | 505.00 (NA) — Standard deviation not calculated because only one participant's sample measured above the assay cut point
  Day 28 | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | 863.00 (NA) — Standard deviation not calculated because only one participant's sample measured above the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | 1493.80 (2.05) | 580.3 (1.15)
  Day 56 | 1461.82 (1.15) | 933.07 (1.16) | 691.90 (1.21) | 1468.22 (1.93) | 1072.06 (1.41)
  Day 84 | 7410.59 (2.59) | 10378.98 (2.87) | 15212.90 (2.54) | 3097.78 (3.24) | 1306.99 (1.01)
  Day 168 | 2578.32 (2.04) | 3554.05 (2.48) | 5344.20 (3.38) | 1901.01 (2.00) | 1241.41 (3.21)
  Day 196 | 24832.80 (3.56) | 32600.15 (3.27) | 48189.54 (2.73) | 12579.63 (5.79) | 2086.94 (1.91)
  Day 280 | 8736.27 (4.24) | 13564.41 (3.06) | 25574.36 (3.65) | 5877.74 (5.45) | 3115.63 (1.35)
  Day 336 | 4977.61 (3.09) | 9543.19 (3.58) | 12351.83 (3.79) | 3719.56 (3.80) | 2907.15 (5.73)

6. Secondary Outcome: Geometric Mean Titer of Antibody Avidity Index Value Against gB
Description: To measure the avidity of responses against CMV gB protein, a standard ELISA assay using recombinant gB protein which did or did not include treatment with 5M urea for 30 minutes of samples after sera had been incubated with recombinant protein. The reported value, or Avidity Index, represents the percent of signal measured in ELISA after treatment with urea relative to samples not exposed to urea.
Time Frame: Through Day 336 or early withdrawal
Population: Analyses were performed on the total vaccinated cohort (TVC), which includes all immunized subjects.
Measure: Geometric Mean (Standard Deviation); unit: Avidity index
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 23 | 26
Avidity index
  Day 28 | 38.98 (1.79) | 41.83 (1.47) | 33.81 (1.52) | 35.53 (2.72) | 38.67 (1.85)
  Day 84 | 64.56 (1.20) | 64.77 (1.22) | 71.91 (1.15) | 57.73 (1.55) | 47.55 (2.10)
  Day 196 | 77.17 (1.14) | 79.58 (1.13) | 83.43 (1.07) | 69.71 (1.29) | 36.39 (2.84)
  Day 336 | 74.82 (1.18) | 75.86 (1.13) | 80.81 (1.09) | 66.43 (1.39) | 44.20 (2.09)

7. Secondary Outcome: Geometric Mean Titer of Neutralizing Antibody Against CMV Infection of Fibroblast Cells
Time Frame: Through Day 196 or early withdrawal
Population: Analyses were performed on the total vaccinated cohort (TVC), which includes all immunized subjects. Samples with antibody titers below the assay cut point were not included in the calculation of geometric mean or standard deviation.
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 23 | 26
Titer
  Day 84 | 77.48 (1.98) | 88.80 (2.19) | 140.38 (2.35) | 107.06 (2.41) | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point
  Day 196 | 139.40 (2.67) | 165.25 (2.29) | 254.31 (2.73) | 101.10 (3.35) | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point

8. Secondary Outcome: Geometric Mean Titer of Neutralizing Antibody Against CMV Infection of Epithelial Cells
Time Frame: Through Day 336 or early withdrawal
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 23 | 26
Titer
  Day 28 | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point
  Day 84 | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | 221.28 (1.57) | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point
  Day 168 | 151.00 (NA) — Standard deviation not calculated because only one participant's sample measured above the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | 177.00 (NA) — Standard deviation not calculated because only one participant's sample measured above the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point
  Day 196 | 159.69 (1.11) | 281.00 (NA) — Standard deviation not calculated because only one participant's sample measured above the assay cut point | 287.24 (1.45) | 261.95 (1.17) | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point
  Day 280 | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | 152.00 (NA) — Standard deviation not calculated because only one participant's sample measured above the assay cut point | 288.17 (1.69) | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point
  Day 336 | 151.00 (NA) — Standard deviation not calculated because only one participant's sample measured above the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | 234.80 (1.82) | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point | NA (NA) — Geometric mean and standard deviation not calculated because all samples measured below the assay cut point

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first injection on Day 0 to Day 336 or early withdrawal, six months post Dose 3 in all participants, in all groups.
Arm/Group | VBI-1501A: 0.5µg With Adjuvant | VBI-1501A: 1.0µg With Adjuvant | VBI-1501A: 2.0 µg With Adjuvant | VBI-1501: 1.0µg Without Adjuvant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 2/26 | 1/26 | 2/25 | 0/26
Other Adverse Events (participants affected / at risk) | 18/25 | 23/26 | 20/26 | 21/25 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VBI-1501A: 0.5µg With Adjuvant (N=25) | VBI-1501A: 1.0µg With Adjuvant (N=26) | VBI-1501A: 2.0 µg With Adjuvant (N=26) | VBI-1501: 1.0µg Without Adjuvant (N=25) | Placebo (N=26)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis Aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VBI-1501A: 0.5µg With Adjuvant (N=25) | VBI-1501A: 1.0µg With Adjuvant (N=26) | VBI-1501A: 2.0 µg With Adjuvant (N=26) | VBI-1501: 1.0µg Without Adjuvant (N=25) | Placebo (N=26)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophageal Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (3) | 1 (2)
Influenza Like Illness (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Malaise (General disorders) | 4 (4) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (15) | 5 (9) | 9 (14) | 6 (8) | 8 (10)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 7 (10) | 2 (2) | 3 (4) | 3 (5)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (9) | 8 (12) | 5 (8) | 6 (6) | 5 (10)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (4) | 2 (2) | 0 (0) | 0 (0)
Orophyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 0 (0) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No